CLINICAL TRIAL: NCT00792610
Title: The Hepatitis B Vaccine Booster Response Among the Youth Who Had Completed Neonatal Hepatitis B Vaccines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: JAN CHYI-FENG/MD, PHD., NATIONAL TAIWAN UNIVERSITY HOSPITAL
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 200701049M; NSC96-2314-B-0020115
Record Dates: First submitted 2008-11-16; First posted 2008-11-18 (Estimated); Results first posted 2009-09-24 (Estimated); Last update posted 2009-10-06 (Estimated); Status verified 2009-08

CONDITIONS: Hepatitis B
Keywords: youth; hepatitis B; vaccination; booster; immunity response
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Vaccines; Engerix-B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hepatitis B booster (Experimental): They receive 3 doses of hepatitis B vaccine (Engerix-B Injection, recombinant HBsAg, 20mcg/ml/vial, GSK) at 0, 1st, 6th month during follow-up. Their anti-HBs status were checked at baseline, one week, one month, sixth month, and seven months later after the first dose of hepatitis B vaccine.
  Interventions: Biological: hepatitis B vaccine

INTERVENTIONS:
Biological: hepatitis B vaccine — Recombinant HBsAg, 20mcg/ml/vial (GSK) one vial IM at Day 0, Month 1, month 6 during follow-up, respectively.
  Other Names: Engerix-B

SUMMARY:
At the time of the present study, the necessity for booster vaccinations for the prevention of hepatitis B(HB) 15 years post-vaccination in the group of young adults who have become seronegative for HB markers after complete neonatal HB vaccination was in question. A booster vaccination strategy may lead to a significant economic impact on national health care resources, and the costs/benefits must therefore be carefully evaluated. Unfortunately, the data to support such analyses are lacking. Because an increased risk of HB infection is anticipated when adolescents enter into young adulthood through becoming sexual active, breakthrough infections such as fulminant HB might be the main concern instead of the risk of chronic HB carriage. To address this issue, this study aimed to measure the booster responses after HB vaccination in seronegative young adults who had completed neonatal HB vaccines in Taiwan before.

DETAILED DESCRIPTION:
This cohort study was conducted between October 2007 and Jan 2009. The target population was subjects aged 18-23 years who were born after 1984 when the Taiwanese national HB vaccination program was launched. Their vaccination records must have shown a completed neonatal HB vaccination, and they were seronegative for all three HB viral markers including HBsAg(Hepatitis B surface antigen), anti-HBc(core antibody against Hepatitis B), and anti-HBs(Surface antibody against Hepatitis B) within 2 years of entry into the study and at study entry. They were recruited through a Student's Health Center Clinic referral, Bulletin Board System posts, and Web-broadcast invitation. The neonatal HB vaccination records were verified through linkage to the Taiwan Center for Disease Control databank. Signed informed consent was obtained from all the participants and their parents or guardians. Pregnant females, persons with a previous history of allergy to HB vaccines, or allergy to yeast were excluded. First 3 months are screen phase to recruit college students for assay of hepatitis B viral markers. Seronegative subjects were approached for enrollment into receiving hepatitis B vaccine booster afterwards.

All participants were tested for HB markers at enrollment, even if they had been tested in the previous months, to confirm their status. A questionnaire was completed at enrolment to record sociodemographic factors including age, gender, self reported family history of hepatitis B carriers, self reported blood type, and so on. The participants then received three intramuscular doses of HB vaccine (Engerix-B, recombinant hepatitis B surface antigen, 20 microgram/ml/vial, GlaxoSmithKline, Belgium) at baseline and at the 1st and 6th month follow-up visits. Their anti-HBs status was checked at baseline, 7-10 days, 1 month, 6 months, and 7 months following the first dose of HB vaccine. Adverse effects associated with the vaccine were also reported within one week after each Engerix-B injection.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-23 years
2. the youth born after July 1984 who have received a hepatitis B virus markers checkup within 2 years including HBsAg, core antibody against hepatitis B(anti-HBc), and surface antibody against hepatitis B (anti-HBs) and the results are all negative for these 3 viral markers.
3. Participants should agree to sign inform consent. For younger than 20 years old subjects, one of their parents also help the participate review and sign the inform consent.
4. Participants are willing to receive 3 doses of Hepatitis B vaccines without payment.
5. General condition is in good health judged by the doctor

Exclusion Criteria:

1. Allergy to Hepatitis B vaccines or yeast
2. pregnancy

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 127 (Actual)
Dates: Start 2007-08; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chyi-Feng Jan, Doctor, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This cohort study was conducted between October 2007 and Jan 2009. The participants were recruited through a Student's Health Center Clinic referral, Bulletin Board System posts, and Web-broadcast invitation. They received intervention and blood exam in the hospital.
Pre-assignment Details: Initially, 150 seronegative subjects for the three hepatitis B viral markers (HBsAg, anti-HBs, and anti-HBc) were invited to participate in the study. Among them, five subjects were excluded because of seropositive results upon recheck or drop-out. History of complete neonatal HB vaccination could not be confirmed in 18 cases.
Period: Overall Study
Arm/Group | Hepatitis B Booster
Started | 127
Youths | 127
Completed | 127
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hepatitis B Booster
Number analyzed (Participants) | 127
Age, Customized [Number; unit: participants]
  < 20 years old | 54
  >= 20 years old | 73
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 66
Blood type [Number; unit: participants]
  A | 28
  B | 31
  AB | 8
  O | 53
  unknown | 7
Body Mass Index(BMI) category [Number; unit: participants] — if BMI< 18.5 then BMIgr3=0; else if BMI >= 18.5 and BMI< 24 then BMIgr3=1; else if BMI >=24 then BMIgr3=2;
  participants
    BMI< 18.5 | 21
    18.5<= BMI < 24 | 94
    BMI >= 24 | 12
Family history of hepatitis B carrier [Number; unit: participants]
  Yes | 18
  NO | 71
  Unknown | 38

OUTCOME MEASURES:

1. Primary Outcome: Hepatitis B Surface Antibody Seroprotective Rate(Seroprotective: for Those Who Had Anti-HBs(Surface Antibody Against Hepatitis B) Titer Higher Than 10 mIU/mL)
Description: The anti-HBs(Surface antibody against Hepatitis B) status was checked at baseline, 7-10 days, 1 month, 6 months, and 7 months following the first dose of hepatitis B vaccine. And then the seroprotective rate for anti-HBs(numbers of those who had anti-HBs titer higher than 10 mIU/mL/all participants numbers) was calculated respectively.
Time Frame: 7 months
Measure: Number; unit: participants
Arm/Group | Hepatitis B Booster
Number analyzed (Participants) | 127
participants
  seroprotective rate of HB vaccine at 7-10 days | 26
  seroprotective rate of HB vaccine at one month | 96
  seroprotective rate of HB vaccine at 6 months | 120
  seroprotective rate of HB vaccine at 7 months | 126
Statistical Analysis 1: Comparison: Hepatitis B Booster; Chi-square analysis and Fischer's exact test were used for comparing group proportions between seropositive and seronegative participants. GMT and their 95% confidence intervals were also calculated using the software developed by Kirkman, T.W. (18) An ANOVA test was performed to compare the difference of the three groups at one, six and seven months categorized by the anti-HBs titers at 7-10 days after the booster; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Risk Difference (RD) = .10, 95% CI [.05 to .15], Standard Deviation .05

ADVERSE EVENTS:
Arm/Group | Hepatitis B Booster
Serious Adverse Events (participants affected / at risk) | 0/127
Other Adverse Events (participants affected / at risk) | 0/127

LIMITATIONS AND CAVEATS:
The possible presence of T cell memory among the seronegative patients for HBsAg(+), anti-HBc(+), and anti-HBs(+) could be a concern.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No